CLINICAL TRIAL: NCT03293043
Title: The University of Alberta Negative Pressure Ventilation Ex-Vivo Lung Perfusion (NPV-EVLP) Trial
Acronym: UA NPV-EVLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00070552
Record Dates: First submitted 2017-09-11; First posted 2017-09-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Ex-Vivo Lung Transplantation

STUDY DESIGN:
Intervention Model Description: The purpose of this Phase I Early Feasibility Proof of Concept clinical trial will be to evaluate initial performance and safety of the NPV-EVLP device to assess and improve the function of marginal donor lungs. By nature, efficacy measures and outcomes of the device will also become evident from the results of this study.
  This is a prospective, non-randomized, interventional trial, taking place solely at the University of Alberta Hospital/Mazankowski Alberta Heart Institute. Lungs deemed marginal, based on standard lung donor criteria that meet the study's eligibility criteria, will be assessed on our NPV-EVLP device to determine suitability for lung transplantation. Objective assessment of quality will be made while the lungs are on the device based on pre-determined functional parameters of lung physiology. Once a total of 12 sets of lungs are transplanted after using the device, safety will be determined by post-operative lung function and recipient survival.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): After initial screening, appropriately obtained informed consent and confirmation of eligibility at time of transplant, those recipients (a total of 12 subjects) who agree to continue as participants will receive reconditioned marginal lungs should the lungs on the device meet acceptable criteria to proceed with clinical transplantation.
  Interventions: Device: NPV-EVLP

INTERVENTIONS:
Device: NPV-EVLP — Lungs deemed marginal based on standard lung donor criteria that meet study eligibility will be physiologically assessed during ex-vivo perfusion. NPV-EVLP of these lungs will be performed with the addition of numerous pre-determined additives. With respect to the decision of lung utilization post-EVLP, eligibility criteria listed in the Post-NPV-EVLP section of the trial will need to be met. Lungs will also be excluded if they are deemed unsuitable based on the clinical judgment of the lung transplant surgeon.

SUMMARY:
This project is focused on helping one of the most vulnerable patient populations in medicine, patients with end-stage chronic lung disease. Lung transplantation is the only cure for end-stage lung disease, however, due to the persistent shortage of donor organs, either due to low organ donation rates or unacceptable organs, only a minority of patients receive desperately needed lung transplants. Currently less than 30% of potential donated thoracic organs are being used for transplantation. The major causes for under utilization of donor thoracic organs are injury sustained by the lungs in trauma or emergency resuscitation or lungs that come from donors who are pronounced dead due to cardiac arrest (known as DCD donors). It has been hypothesized that these injuries may be reversible or repairable if there was an opportunity to evaluate and repair these organs outside of the body (ex-vivo), prior to transplantation. In fact, studies have shown that the use of normothermic Ex-Vivo Lung Perfusion (EVLP) has increased the rate of donor organ utilization at centers that have adopted the technology.

Current methodology for all clinically available EVLP devices uses Positive Pressure Ventilation (PPV). Researchers at the University of Alberta (UofA), however, have developed an EVLP device that will apply Negative Pressure Ventilation (NPV) to the lungs, as opposed to PPV, which is the most ideal mimicry of native lung physiology. The objective of this early feasibility safety trial is to show that the UofA developed NPV-EVLP device is acceptable in evaluating and improving the quality of marginal donor lungs compared to currently used EVLP devices, ultimately allowing for these types of donor lungs to be safely transplanted into patients on the lung transplant recipient waitlist.

ELIGIBILITY:
5.2 PRE-NPV-EVLP Donor Eligibility Criteria

5.2.1 Donor MUST meet ANY ONE of the following Inclusion Criteria to proceed with NPV-EVLP:

1. Best ratio of the PaO2 to FiO2 of < 300mmHg;
2. Pulmonary edema, defined as bilateral interstitial infiltrates without evidence of infection, detected on the last chest radiograph by the lung-transplantation physician assessing the donor;
3. Poor lung deflation or inflation during direct intraoperative visual examination at the donor site;
4. Donor age is ≥ 55 years;
5. Expected cold ischemic time > 6 hours;
6. Blood transfusions ≥ 10 units; or
7. Donation after cardiac death (DCD), as defined by Maastricht category III (donor without a heartbeat and with cardiocirculatory death imminent after withdrawal of treatment) or category IV (cardiocirculatory death in a brain-dead donor).

5.2.2 Donor Exclusion Criteria to NOT proceed with NPV-EVLP:

1. Donor lungs with established pneumonia;
2. Severe mechanical lung injury (i.e., contusions in more than one lobe) or trauma determined by chest x-ray, bronchoscopy, CT scan or visual inspection; or
3. Gross gastric aspiration within the lungs
4. Donor lungs have active infectious disease such as HIV, Hepatitis B, Hepatitis C, West Nile Virus (WNV), HTLV, or Syphillis (if this information not available at start of EVLP, it should be re-assessed prior to transplant).

5.3 POST-NPV-EVLP Donor Eligibility Criteria

5.3.1 Donor Inclusion Criteria to proceed with Transplant:

1. Surgeon must be satisfied with the clinical evaluation and appearance of the lungs; if not, reason for refusal must be documented;
2. Lungs show PaO2/FiO2 ratio ≥ 350mmHg; AND
3. Deterioration of less than 15% from baseline for physiological measurements pulmonary vascular resistance (PVR), dynamic compliance and peak inspiratory pressure.

5.3.2 Donor Exclusion Criteria to proceed with Transplant:

1. Lungs show a PaO2/FiO2 ratio of < 350mmHg;
2. Greater than 15% functional deterioration across the following physiological parameters: PVR, dynamic compliance and peak inspiratory pressure;
3. Donor lungs are positive for infectious disease such as HIV, Hepatitis B, Hepatitis C, West Nile Virus (WNV),HTLV, or Syphillis.

5.4 Recipient Eligibility Criteria

5.4.1 Recipient Inclusion Criteria

1. Patients on our institution's waitlist requiring bilateral transplantation
2. Male or Female 18 years of age or older
3. Written informed consent provided.

5.4.2Recipient Exclusion Criteria

1. Multi-organ recipient or re-transplant
2. HIV, Hepatitis, or other infection that excludes subject from transplant in the study
3. Subject is on hemodialysis or has chronic severe renal dysfunction
4. Concurrent cardiac procedure
5. Recipient is on Nova Lung, ECMO or on mechanical ventilation (CPAP and BiPAP not exclusionary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Patient survival post transplantation at Day30 | Day30 post-Transplant
  The primary end point is a co-primary endpoint comparing patient survival rates post transplantation at Day30 (Outcome 1) and rates of Primary Graft Dysfunction (PGD) Grade 3 in the first 72 hours (Outcome 2) with success measured only if both endpoints are met.
Primary Graft Dysfunction (PGD) Grade 3 in the first 72Hours | First 72Hours post-Transplant
  The primary end point is a co-primary endpoint comparing patient survival rates post transplantation at Day30 (Outcome 1) and rates of Primary Graft Dysfunction (PGD) Grade 3 in the first 72 hours (Outcome 2) with success measured only if both endpoints are met.

SECONDARY OUTCOMES:
Primary Graft Dysfunction (PGD) Grades | Time0 (ICU Admission), Time24Hours (post-Transplant), Time48Hours (post-Transplant), and Time72Hours (post-Transplant)
  PGD scores will be assessed a Grade of 0, 1, 2 or 3 (per ISHLT Guidelines) at Time0 (ICU Admission), Time24Hours (post-Transplant), Time48Hours (post-Transplant), and Time72Hours (post-Transplant) with respect to PaO2/FiO2 ratios and presence/absence of radiographic infiltrates consistent with pulmonary edema.
ICU LOS | From admission to the ICU through to exact date of ICU Discharge (up to 30Days)
  ICU length of stay (LOS) post-Transplant will be captured.
Hospital LOS | From date of Transplant through to exact date of Index Hospital Discharge (up to 6Months)
  Index hospital length of stay (LOS) length of stay post-Transplant will be captured until D/C.
Duration of Mechanical Ventilation post-Transplant | Time0 (ICU Admission post-Transplant) through to exact time of extubation post-Transplant
  The duration of Mechanical Ventilation post-Transplant will be captured until extubation.
FEV1 | 6Months and 1Year
  FEV1 results from spirometry efforts at 6Months and 1Year will be captured.
Quality of Life (SF-36) | 6Months and 1Year
  Quality of Life measured by the 36-Item Short Form Survey (SF-36) at 6Months and 1Year will be captured.

OTHER OUTCOMES:
Safety endpoints as defined by the number of lung-related serious adverse events (SAEs) to Day30 | To Day30 post-Transplant
  Safety endpoints include the number of lung-related serious adverse events (SAEs) through to the Day30 follow-up after transplantation (T0) per subject. This endpoint will be defined to consist of the following serious adverse events: Acute rejection, Respiratory failure, Bronchial anastomotic complication, and Major pulmonary-related infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jayan Nagendran, MD, PhD, Principal Investigator — Cardiac Surgeon, Director of Research, Associate Professor, University of Alberta; Darren Freed, MD, PhD, Principal Investigator — Cardiac Surgeon, Associate Professor, University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Only aggregate and descriptive data of the experimental group vs the SOC arm will be shared in the form of publications.

REFERENCES:
- [Derived] Buchko MT, Boroumand N, Cheng JC, Hirji A, Halloran K, Freed DH, Nagendran J. Clinical transplantation using negative pressure ventilation ex situ lung perfusion with extended criteria donor lungs. Nat Commun. 2020 Nov 13;11(1):5765. doi: 10.1038/s41467-020-19581-4. PMID 33188221